CLINICAL TRIAL: NCT02081625
Title: Exploratory Study of NS-065/NCNP-01 in Duchenne Muscular Dystrophy
Brief Title: Exploratory Study of NS-065/NCNP-01 in DMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCNP/DMT01; UMIN000010964 (Other: UMIN-CTR)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; NS-065/NCNP-01; exon 53 skipping; morpholino
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NS-065/NCNP-01 (Experimental)
  Interventions: Drug: NS-065/NCNP-01

INTERVENTIONS:
Drug: NS-065/NCNP-01 — NS-065/NCNP-01 for Infusion is packaged as 25 mg/mL in phosphate buffered saline with 1 mL per vial. Study dosages will be infused over a 1 hour period with Normal saline as follows:
  Cohort 1: 1.25mg/kg once weekly for 12 weeks; Cohort 2: 5.0mg/kg once weekly for 12 weeks; Cohort 3: 20.0mg/kg once weekly for 12 weeks

SUMMARY:
This study is designed to assess the safety, tolerability, efficacy and pharmacokinetics (PK) of NS-065/NCNP-01 in subjects diagnosed with Duchenne muscular dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

Subject with Duchenne muscular dystrophy eligible for enrolment in the study must meet all of the following criteria:

1. Has an out of frame deletion(s) that could be corrected by skipping exon 53 as confirmed by any of methodology at the time of visit 1. If not confirmed by any of methodology that evaluates the relative copy number of all exons (i.e. MLPA, CGH etc), must be confirmed through these techniques by the time of visit 4.
2. DNA sequencing of exon 53 confirms that no DNA polymorphisms occur that could compromise duplex formation between NS-065/NCNP-01 and pre-mRNA.
3. There is confirmation of detection of dystrophin mRNA with skipping of exon 53 and dystrophin production after in vitro exposure of NS-065/NCNP-01 to subject-derived cells.
4. Male and >= 5 years and < 18 years of age at the time of obtaining informed consent and/or assent.
5. Able to give informed consent in writing signed by parent(s) or legal guardian who is able to understand all of the study procedure requirements. If applicable, able to give informed assent in writing signed by the subject.
6. Life expectancy of at least 1 year
7. Unable to ambulate. Ambulant subject can be enrolled according to the circumstances.
8. Have intact muscles, which have adequate quality for biopsy. (No lacks or severe atrophy of tibialis anterior muscle)
9. QTc <450 msec (based on 12-lead ECGs), or <480 msec for subject with Bundle Branch Block.
10. If taking glucocorticosteroids, no significant change in total daily dosage or dosing regimen after the time of visit 1.

Exclusion Criteria:

Subject with Duchenne muscular dystrophy meeting any of the following criteria must not be enrolled in the study:

1. Has participated in other pharmacological clinical trial that might recover dystrophin protein by the readthrough or the exon-skipping therapy, and/or upregulate the dystrophin-associated proteins such as utrophin.
2. A forced vital capacity (FVC) < 50% of predicted.
3. A left ventricular ejection fraction (EF) < 40% or fractional shortening (FS) < 25% based on echocardiogram (ECHO).
4. Surgery within the last 3 months prior to the first anticipated administration of study medication or planned for anytime during the duration of the study.
5. Positive hepatitis B surface antigen (HbsAg), hepatitis C antibody test (HCV), or human immunodeficiency virus (HIV) test at screening.
6. Current diagnosis of any immune deficiency or autoimmune disease.
7. Current diagnosis of any active or uncontrolled infection, cardiomyopathy, or liver or renal disease.
8. Use of any other investigational agents and/or experimental agents within 3 months prior to the first anticipated administration of study medication.
9. History of any severe drug allergy.
10. Unable to give informed consent about using adequate contraception from the first administration until at least 6 months after the last dose of study medication, by parent(s) or legal guardian.
11. Subject considered by the investigator (or sub-investigator), for any reason, to be an unsuitable candidate for the study.

    -

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse event and adverse drug reaction) | Up to 15-17 weeks (12 weeks treatment period and 3-5 weeks follow up period)

SECONDARY OUTCOMES:
Expression of dystrophin protein | At 14-15 weeks (2-3 week after from 12 weeks treatment period)
Detection of exon53 skipped mRNA of dystrophin | At 14-15 weeks (2-3 week after from 12 weeks treatment period)
NS-065/NCNP-01 concentration of the blood plasma | 12 weeks
NS-065/NCNP-01 concentration of the urine | 12 weeks
Serum Creatine kinase concentration | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shin'ichi Takeda, MD, PhD, Study Director — National center of Neurology and Psychiatry; Hirofumi Komaki, MD, PhD, Principal Investigator — National center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan